CLINICAL TRIAL: NCT02425046
Title: Family Obesity Intervention: Motivational Interviewing and Community Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helena Laroche (Other)
Responsible Party: Sponsor-Investigator, Helena Laroche, Physician, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201406722
Record Dates: First submitted 2014-12-11; First posted 2015-04-23 (Estimated); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: family
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- health coaching and community screening (Experimental): Family Health Coaching and community benefits screening
  Interventions: Behavioral: health coaching; Behavioral: community screening
- community screening (Other): community benefits screening only
  Interventions: Behavioral: community screening

INTERVENTIONS:
Behavioral: health coaching — Health coaching using motivational interviewing focus on family diet and exercise change and connection with community resources specific to goals set.
  Arms: health coaching and community screening
Behavioral: community screening — Screening for community resources that families may be eligible for to receive help with basic needs including shelter, food, health insurance etc.

SUMMARY:
Low-income children and children of obese parents are at high risk of obesity. Effective interventions are needed to target these families to improve the health of the parents and prevent obesity in the children. The hypothesis is that an intervention that combines engagement of community organizations, motivational interviewing (MI, a technique proven to help people set goals that are personally meaningful), and resource mobilization will change diet and physical activity habits among disadvantaged families. This proposal grew from an established community-based participatory research (CBPR) partnership between the research team and community organizations that serve high minority (45-55%), low-income populations. Partners include a community health center, a food pantry network, a work-force training program, and other agencies. These partners designed and implemented a successful pilot project on which this proposal is based. The specific aims of this proposal are 1) To evaluate the efficacy of a family-targeted obesity intervention based on MI and resource-mobilization. Hypotheses: In comparison to control families, families participating in the intervention will demonstrate a) a reduction in BMI for adults, b) an increase in minutes of moderate physical activity and decreased sedentary time for both adults and children accelerometer), and c) a reduction in the number of obesity risk behaviors and an increase in obesity prevention behaviors among children. 2) To examine the mediators of intervention effects. 3) Identify the types of resources needed most often by intervention families to support lifestyle change. This randomized controlled trial includes 260 low-income families that contain at least one obese adult and one normal or overweight child between 6 and 12. The 12-month intervention has two elements. 1) A health coach will use MI to help families explore ambivalence toward and motivations for change and set goals for improving diet and physical activity. 2) To support goals, families will be connected with community agencies that can assist with general (e.g., financial) and goal specific resources (e.g., food, physical activity opportunities). Collaboration between organizations will streamline referrals, maximize resources, and facilitate access. Control families will get a basic screen for needs and information about available community resources. Outcomes are measured at baseline, 6, 12, and 18 months. This intervention is innovative in that it 1) focuses on lifestyle changes for the entire family and measures outcomes in adults and children, 2) combines MI focused on the entire family and community resource referrals specific to family needs and goals for change, 3) partners community organizations to coordinate resources for families, and 4) involves partners in all research phases via a CBPR approach. This contribution will be significant because the proposed intervention, if successful, can be replicated elsewhere and adapted to the local resource environment to address adult obesity and prevent childhood obesity in a high-risk population. The study will also identify the types of resources low-income families need to change diet and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* one parent must have a BMI of 30 or above, and be parent or guardian of at least one child
* between the ages of 6 and 12. Children this age are targeted because they benefit most from parental involvement
* are old enough to participate in family goal setting and activities, but young enough to be heavily influenced by family environment.
* a child must live with the obese parent at least 80% of the time.

Exclusion Criteria:

* adults with obesity or target children with a medical condition or medication that significantly alters their

  1. ability to follow the dietary recommendations (e.g., renal diet, severe food allergy, celiac disease)
  2. mobility (e.g. bed bound or unable to participate in any sort of physical activity even with assistive devices), or
  3. weight
* additionally we will exclude those who have a significant psychiatric disease, substance abuse disorder or cognitive impairment that would interfere with their ability to participate
* those with controlled or mild depression would not be excluded
* adults with hypertension, type II diabetes, or glucose intolerance will not be excluded, as advocated changes are consistent with their needs
* no data will be collected from non-target children who meet the exclusion criteria.
* adults with obesity who are currently pregnant at baseline will be excluded because of their altered weight and dietary patterns. If the adult with obesity becomes pregnant during the intervention their family will be allowed to continue in the intervention but the pregnant adults' anthropometric data will not be collected.
* the intervention will intentionally target low-income families through recruitment site choices but will not exclude or include families based on income requirements.
* pregnant women will not be targeted but may be included if not the adult with obesity (see above).
* weight, height, waist circumference will not be collected on pregnant women.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: helena Laroche, MD, Principal Investigator — University of Iowa
Locations (3):
- United States (3):
  - Primary Health Care, Inc, Des Moines, Iowa
  - DMARC food pantries, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: Yes
Investigator will contact PI to discuss their interest in using the data to learn about what is available - data dictionary (code book) of variable names may be made available. Investigator must complete a form outlining what analysis they are proposing. Investigator must sign a confidentiality agreement. Data provided in de-identified format and must be destroyed after analysis and publication is complete.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available after 18-month data has been processed and cleaned. Estimated date: June 2020 (subject to change, dependent on COVID-19).
Access Criteria: Form will be reviewed by the PI, University of Iowa investigative team and the community advisory board and a decision about approval will be made. A University of Iowa research team member must be included in the analysis team to help with context and interpretation of data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After baseline data collection, participants were not randomized until the were able to be contacted by phone by the community resource specialist who explained the randomization process again and provided them with their assignment. If participants were no longer able to be contacted or no longer wished to participate after baseline data collection they were not randomized.
  Numbers reflect the total number of unique participants and not the number of dyads.
Groups:
- Health Coaching and Community Screening: Family Health Coaching and community benefits screening
  health coaching: Health coaching using motivational interviewing focus on family diet and exercise change and connection with community resources specific to goals set.
  community screening: Screening for community resources that families may be eligible for to receive help with basic needs including shelter, food, health insurance etc.
  Written information on healthy family diet and exercise
- Community Screening: community benefits screening only
  community screening: Screening for community resources that families may be eligible for to receive help with basic needs including shelter, food, health insurance etc.
  Written information on healthy family diet and exercise
- Lost to Follow up Before Randomization: Participants unable to be contacted after baseline and thus never randomized to an intervention group per protocol.
Period: Overall Study
Arm/Group | Health Coaching and Community Screening | Community Screening | Lost to Follow up Before Randomization
Started | 206 | 210 | 56
Completed | 138 | 148 | 0
Not Completed | 68 | 62 | 56
Not completed — Lost to Follow-up | 52 | 50 | 56
Not completed — Withdrawal by Subject | 16 | 12 | 0

BASELINE CHARACTERISTICS:
Population: A total of 208 adult-child pairs (416 participants) were randomized - baseline information is provided on them. The 28 adult-child pairs (56 participants) who were consented but who were not randomized (per protocol because of loss to follow up) are not included in these numbers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Coaching and Community Screening | Community Screening | Total
Number analyzed (Participants) | 103 | 105 | 208
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Adult | 35.1 (7.1) | 35.2 (7.1) | 35.1 (7.2)
  Child | 8.4 (2.0) | 8.8 (2.0) | 8.6 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Adult: Female | 98 | 100 | 198
  Adult: Male | 5 | 5 | 10
  Child: Female | 48 | 52 | 100
  Child: Male | 55 | 53 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Adult: Hispanic or Latino | 25 | 31 | 56
  Adult: Not Hispanic or Latino | 77 | 74 | 151
  Adult: Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Adult: American Indian or Alaska Native | 0 | 0 | 0
  Adult: Asian | 0 | 0 | 0
  Adult: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Adult: Black or African American | 32 | 34 | 66
  Adult: White | 43 | 42 | 85
  Adult: More than one race | 0 | 0 | 0
  Adult: Unknown or Not Reported | 28 | 29 | 57
  Child: American Indian or Alaska Native | 0 | 0 | 0
  Child: Asian | 0 | 0 | 0
  Child: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Child: Black or African American | 31 | 34 | 65
  Child: White | 47 | 48 | 95
  Child: More than one race | 0 | 0 | 0
  Child: Unknown or Not Reported | 25 | 23 | 48
Education Level, Adults [Count of Participants; unit: Participants]
  High School Not Completed | 27 | 26 | 53
  High School Graduate | 51 | 51 | 102
  College Graduate | 24 | 28 | 52
  Unknown | 1 | 0 | 1
Diabetes Status (Adults) [Count of Participants; unit: Participants]
  Diabetes | 8 | 8 | 16
  Prediabetes | 5 | 9 | 14
  Neither | 87 | 86 | 173
  Unknown | 3 | 2 | 5
Family Income (before taxes), Adults [Mean (Standard Deviation); unit: dollars] | 29987 (29503) | 26979 (24818) | 28437 (26189)
BMI, kg/m^2, Adults [Mean (Standard Deviation); unit: kg/m^2] | 39.1 (7.1) | 39.7 (7.2) | 39.4 (7.35)
BMI z-score (BMIz), Child [Mean (Standard Deviation); unit: BMI z-score (BMIz)] — The BMI z-score (BMIz) indicates the number of standard deviations away from the mean BMI for age and sex as determined by the CDC growth curves. A z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
  BMI z-score (BMIz) | 1.2 (1.0) | 1.1 (1.0) | 1.1 (1.1)
Family Nutrition and Physical Activity Scale, Child [Mean (Standard Deviation); unit: Unit on a scale] — The Family Nutrition and Physical Activity Scale is a 20 item measure of family behaviors linked to childhood obesity either as protective behaviors or behaviors that promote obesity. Each question may contribute a score between from 1 to 4. Thus the potential score ranges from 20 to 80 and a higher score reflects fewer behaviors thought to contribute to obesity and more behaviors beneficial to obesity prevention.
  Unit on a scale | 60.1 (8.1) | 59.6 (9.2) | 59.8 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Adult Body Mass Index
Description: Change in Adult BMI from baseline to 12 months
Time Frame: Outcome was assessed at baseline and 12 months and then calculated by subtracting the baseline value from the value at 12 months
Population: All adult participants who were randomized.
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Health Coaching and Community Screening | Community Screening
Number analyzed (Participants) | 103 | 105
kg/m2 | 0.3 (0.9) | -0.1 (0.7)
Statistical Analysis 1: Comparison: Health Coaching and Community Screening vs Community Screening; Test type: Superiority; p = 0.67, t-test, 2 sided — Threshold for statistical significance <0.05; Multiple imputation used to fill in missing data - imputation included demographic and 6 month data. 5 datasets created and results averaged

2. Primary Outcome: Change From Baseline in Duration of Daily Moderate to Vigorous Physical Activity
Description: Moderate to vigorous physical activity of the target adult measure by an accelerometer at baseline and 12 months. Calculated by subtracting the baseline amount from the 12 month value. The accelerometer is a wrist worn device - worn for 7 days - which measures motion in three directions - the amount of motion is then used assess what level of physical activity the participant is doing at each time interval. Vigorous - such as running, moderate such as fast walking, light such as walking slowly.
Time Frame: measured at baseline and 12 months - outcome is the change from baseline to 12 months.
Population: All target adults randomized
Measure: Mean (Standard Error); unit: minutes per day
Arm/Group | Health Coaching and Community Screening | Community Screening
Number analyzed (Participants) | 103 | 105
minutes per day | -2.7 (9.0) | 0.5 (5.2)
Statistical Analysis 1: Comparison: Health Coaching and Community Screening vs Community Screening; null hypothesis - there will be no difference between the groups; Test type: Superiority; p = 0.735, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Change in Score for Target Child Over 12months on the Family Nutrition and Physical Activity Scale
Description: Change in the Family Nutrition and Physical Activity Scale from baseline to 12 months - measure of behaviors relate to childhood obesity - parent reports for the target child. Scale scores possible range from 20 to 80. Higher indicates healthier behaviors.
Time Frame: measured at baseline and 12 months
Population: All target children randomized
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Health Coaching and Community Screening | Community Screening
Number analyzed (Participants) | 103 | 105
units on a scale | 2.2 (0.9) | 2.8 (1.0)
Statistical Analysis 1: Comparison: Health Coaching and Community Screening vs Community Screening; Null hypothesis that there would be no difference in change in FNPA scores between the two groups over 12 months; Test type: Superiority; p = 0.599, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]

4. Primary Outcome: Target Child - Change in Daily Moderate to Vigorous Physical Activity
Description: Change in minutes per day of moderate to vigorous physical activity of the target child as measure by accelerometer from baseline to 12 months. Calculated by subtracting the baseline amount from the 12 month value. The accelerometer is a wrist worn device - worn for 7 days - which measures motion in three directions - the amount of motion is then used assess what level of physical activity the participant is doing at each time interval. Vigorous - such as running, moderate such as fast walking, light such as walking slowly.
Time Frame: baseline and 12 months
Population: All target children randomized
Measure: Mean (Standard Error); unit: minutes per day
Arm/Group | Health Coaching and Community Screening | Community Screening
Number analyzed (Participants) | 103 | 105
minutes per day | -7.0 (3.0) | -9.6 (3.3)
Statistical Analysis 1: Comparison: Health Coaching and Community Screening vs Community Screening; Null hypothesis: Change in MVPA from baseline to 12 months will not be different between target children in the two groups; Test type: Superiority; p = 0.583, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Adult - Change From Baseline in Number of 12 Ounce Cups or Cans Per Day of Sugar Sweetened Beverages
Description: Change in self-reported sugar-sweetened beverage intake per day from baseline to 12 months as reported by participant in numbers of 12 ounce cups or cans.
Time Frame: baseline and 12 months
Population: All randomized target adults
Measure: Mean (Standard Error); unit: # of 12 ounce cups per day
Arm/Group | Health Coaching and Community Screening | Community Screening
Number analyzed (Participants) | 103 | 105
# of 12 ounce cups per day | -0.6 (0.4) | -1.3 (0.4)
Statistical Analysis 1: Comparison: Health Coaching and Community Screening vs Community Screening; Null hypothesis is that there will be no difference between the two arms in change in sugar sweetened beverage intake over 12 months; Test type: Superiority; p = 0.312, t-test, 2 sided; Multiple imputation including demographics and 6 month data used to complete dataset. 5 datasets created and t-score averaged

6. Secondary Outcome: Adult - Physical Activity Questionnaires:
Description: Reported leisure activity time on the Global Physical Activity Questionnaire reported in minutes per day.
Time Frame: 12 month
Population: All randomized target adult participant who completed the GPAQ questionnaire. One participant removed for implausible value at baseline. Linear Mixed Models used all participants.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Health Coaching and Community Screening | Community Screening
Number analyzed (Participants) | 102 | 105
minutes per day | 120 (188) | 100 (193)
Statistical Analysis 1: Comparison: Health Coaching and Community Screening vs Community Screening; Linear quantile mixed models (a non-parametric linear mixed model) was used because because of non-normal distribution that could not be remedied by transformation; Test type: Superiority; p = 0.10, Linear quantile mixed model; Linear quantile mixed models (a non-parametric linear mixed model) was used because of non-normal distribution that could not be transformed; difference in change between two arms = 75, 95% CI 2-sided [-15 to 165] — Comparison of the intervention target adult change in reported physical activity compared to the control group

7. Secondary Outcome: Adult - Waist Circumference:
Description: waist circumference in centimeters
Time Frame: 12 months
Population: Every randomized participant with a valid waist circumference measurements at baseline was used in statistical analysis. For means reported below only those with data at 12 months are used 68 control and 65 intervention.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Health Coaching and Community Screening | Community Screening
Number analyzed (Participants) | 65 | 68
centimeters | 114.3 (13.8) | 119.7 (14.9)
Statistical Analysis 1: Comparison: Health Coaching and Community Screening vs Community Screening; Test type: Superiority; p = 0.057, Mixed Models Analysis; difference in change between two arms = -2.54, 95% CI 2-sided [-5.14 to 0.07] — The intervention arm in comparison to the control arm

8. Secondary Outcome: Child - BMI Z-score:
Description: Change in child BMI z-score from baseline to 12 months. The BMI z-score (BMIz) indicates the number of standard deviations away from the mean BMI for age and sex as determined by the CDC growth curves. A z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: 12 months
Population: All target children randomized
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Health Coaching and Community Screening | Community Screening
Number analyzed (Participants) | 103 | 105
units on a scale | 0.0 (0.04) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Health Coaching and Community Screening vs Community Screening; Test type: Superiority; p = 0.874, t-test, 2 sided; [statistical method as in outcome 5, analysis 1]

9. Secondary Outcome: Child - Screen Time Questionnaire:
Description: total hours of screen time per week as collected by questionnaire given to the parent
Time Frame: 12 months
Population: Randomized target/Index Child whose parents completed the screen time questionnaire at baseline. All data used for LQMM model. Means provided based only on those who completed the 12 month questionnaire - 71 control and 67 intervention
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Health Coaching and Community Screening | Community Screening
Number analyzed (Participants) | 67 | 71
hours per week | 27 (12.9) | 29 (12.3)
Statistical Analysis 1: Comparison: Health Coaching and Community Screening vs Community Screening; Test type: Superiority; p = 0.31, Mixed Models Analysis; Screen time was log transformed to normalized the distribution. Results have been back transformed from log 10 scale; % difference in change between arms = 7, 95% CI 2-sided [-7 to 23] — % change in screen time of the intervention arm compared to the control arm

10. Secondary Outcome: Child -Dietary Measures: Change in 12 Ounce Cups Per Day of Sugar Sweetened Beverages
Description: Change in parent reported sugar-sweetened beverage intake per day from baseline to 12 months as reported per 12 ounce cup or can. Calculate by subtracting the baseline value from the 12 month value.
Time Frame: baseline and 12 months
Population: All targeted children randomized
Measure: Mean (Standard Error); unit: # of 12 ounce cups per day
Arm/Group | Health Coaching and Community Screening | Community Screening
Number analyzed (Participants) | 103 | 105
# of 12 ounce cups per day | -0.5 (0.2) | -0.7 (0.3)
Statistical Analysis 1: Comparison: Health Coaching and Community Screening vs Community Screening; Test type: Superiority; p = 0.516, t-test, 2 sided; [statistical method as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Health Coaching and Community Screening | Community Screening
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/105
Other Adverse Events (participants affected / at risk) | 0/103 | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT02425046/Prot_SAP_000.pdf